CLINICAL TRIAL: NCT00535145
Title: A Single-arm Evaluation of the Safety of Paliperidone Extended-Release (ER) in Subjects With Schizophrenia or Schizoaffective Disorder With Hepatic Disease
Brief Title: Study to Measure the Safety of Paliperidone ER (Extended-release) in Patients With Liver Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014341; R076477SCH4005 (Other: Ortho McNeil Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2013-09-20 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychotic Disorders
Keywords: antipsychotic; paliperidone ER; liver disease; Schizophrenia; Schizoaffective Disorder; Invega
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Liver Diseases | interventions — Therapeutics; Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Treatment as usual (TAU), Paliperidone ERTreatment as usual is the subject's current antipsychotic and doses for 4 weeks; TAU AND Paliperidone ER - per site investigator for 1 week; Paliperidone ER 6mg once daily for 1 week; Paliperidone ER-3 to 12mg tablets once daily for 4 weeks
  Interventions: Drug: Treatment as usual (TAU), Paliperidone ER

INTERVENTIONS:
Drug: Treatment as usual (TAU), Paliperidone ER — Treatment as usual is the subject's current antipsychotic and doses for 4 weeks; TAU AND Paliperidone ER - per site investigator for 1 week; Paliperidone ER 6mg once daily for 1 week; Paliperidone ER-3 to 12mg tablets once daily for 4 weeks

SUMMARY:
The purpose of this study is to evaluate the tolerability and safety of paliperidone ER (extended-release) in doses between 3 milligrams per day and 12 milligrams per day in the treatment of patients with schizophrenia or schizoaffective disorder and liver disease.

DETAILED DESCRIPTION:
Patients with schizophrenia or schizoaffective disorder commonly have other conditions that may affect the liver, such as alcohol abuse and/or chronic liver infections (hepatitis). Although single-dose studies in patients with liver disease are conducted to test the safety of medications, there is less information about the safety of treatment with medications for schizophrenia in this at-risk population of patients with schizophrenia or schizoaffective disorder and liver disease. This 9-week study is open-label (both patient and investigators know what study drug and dose of study drug the patient is taking) and has 2 phases. During Phase 1, which lasts 4 weeks, patients will continue to take whatever medication they are already taking for schizophrenia (TAU, or treatment as usual). During the first week of Phase 2, patients will receive decreasing doses of TAU and increasing doses of paliperidone ER. For the rest of Phase 2, which lasts 4 more weeks, patients will take paliperidone ER in doses between 3 mg/day and 12 mg/day, as prescribed by the study doctor. This study will evaluate adverse events and will use several scales and tests to measure the effectiveness of paliperidone ER in patients with an established diagnosis of schizophrenia or schizoaffective disorder and liver disease. Study assessments include the PANSS (Positive and Negative Symptom Scale for Schizophrenia), CGI (Clinical Global Impression scale), MSQ (Medication Satisfaction Questionnaire), sleep VAS (Visual Analog Scale), SF-36 (Short Form 36 Health Survey), and PSP (Personal and Social Performance Scale). Each assessment will be performed at least two times during the course of the study, but some assessments will be done more frequently. Visits are scheduled every 1 to two weeks during the 9 week study.

The hypothesis is that paliperidone ER can be used safely in patients with schizophrenia or schizoaffective disorder who also have identified liver disease. During Phase 1 of the study, patients will continue to take whatever medication they are already taking for schizophrenia (TAU, or treatment as usual) for 4 weeks. For the first week of Phase 2, patients will receive decreasing doses of TAU. During Phase 2, patients will take paliperidone ER in doses between 3 milligrams per day and 12 milligrams per day by mouth for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal for at least 1 year, surgically sterile, abstinent, or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study, and must also have a negative urine pregnancy test at Screening
* Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) diagnosis of schizophrenia or schizoaffective disorder
* Must have identified current, stable liver disease (e.g., viral hepatitis, alcoholic cirrhosis)
* Child-Pugh class A or B (total score < 10)

Exclusion Criteria:

* Not able to swallow the study medication whole with the aid of water
* Not currently meeting criteria for any other Axis I diagnosis, including a DSM-IV diagnosis of Bipolar Disorder
* Not using alcohol in the previous 2 weeks or meeting the DSM-IV criteria for substance abuse or dependence or alcohol abuse or dependence in the 6 months before study entry
* Not experiencing severe liver disease or an acute exacerbation of the underlying liver disease (Child-Pugh total score >=10)
* No evidence of severe hepatic decompensation within the previous 3 months, such as: ascites not controlled with diuretics, peritonitis, portal hypertension or gross hepatic encephalopathy (eg, somnolence, stupor, coma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC
Locations (21):
- United States (21):
  - Cerritos, California
  - Chino, California
  - Garden Grove, California
  - Huntington Beach, California
  - Santa Ana, California
  - Torrance, California
  - Fort Lauderdale, Florida
  - Hollywood, Florida
  - Kissimmee, Florida
  - Lake Charles, Louisiana
  - Flowood, Mississippi
  - Kansas City, Missouri
  - Clementon, New Jersey
  - Albuquerque, New Mexico
  - Staten Island, New York
  - Cincinnati, Ohio
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Sioux Falls, South Dakota
  - Irving, Texas
  - White River Junction, Vermont

REFERENCES:
- See also: A Single-Arm Evaluation of the Safety of Paliperidone Extended-Release (ER) in Subjects with Schizophrenia or Schizoaffective Disorder with Hepatic Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=942&filename=CR014341_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One-hundred-twenty-one (121) participants were enrolled but only 114 entered Phase 1 of the study (5 participants enrolled twice and only had their first entrance included and 2 participants did not sign the required HIPAA form).
Groups:
- Study Treatment: Phase 1; Day 1 through Day 27: Patients took therapy for schizophrenia as prescribed before study entry (referred to "treatment as usual" abbreviated as "TAU") for 4 weeks. Phase 2; Day 28 through Day 62: The dose of TAU was then tapered (reduced and stopped) over a 1-week period and treatment started with paliperidone extended-release (ER) tablets, 6 mg, orally (by mouth) once daily followed by 4 weeks of paliperidone ER, 3-12 mg once daily as monotherapy (treatment with Paliperidone ER alone)
Period: Phase I
Arm/Group | Study Treatment
Started | 114
Completed | 85
Not Completed | 29
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 6
Not completed — (eligibility) | 8
Not completed — (protocol violation) | 1
Not completed — (PI decision) | 1
Not completed — (diagnosis) | 3
Period: Phase II
Arm/Group | Study Treatment
Started | 84 (Of the 85 participants who completed Phase 1, 84 met the criteria to enroll into Phase 2)
Completed | 69
Not Completed | 15
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 5
Not completed — Subject non-compliance | 2

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 57

OUTCOME MEASURES:

1. Secondary Outcome: Positive and Negative Symptoms of Schizophrenia (PANSS) Change From Baseline
Description: The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale (1="Absent", 2="Minimal", 3="Mild", 4="Moderate", 5="Moderate/Severe", 6="Severe", 7="Extreme").The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate more severe neuropsychiatric symptoms of schizophrenia.
Time Frame: Day 1 - Day 62
Population: Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Study Treatment: Day 1 through Day 27: Antipsychotic treatment as usual (TAU); Day 28 through Day 62: Paliperidone ER (1 week cross titration plus 4 weeks mono-therapy).
Arm/Group | Study Treatment
Number analyzed (Participants) | 79
Scores on a scale
  Day 27 (n=79) | -1.7 (7.35)
  Day 48 (n=74) | -5.4 (8.72)
  Day 62 (n=77) | -7.2 (9.91)
  Post Day 27 Endpoint (n=79) | -7.6 (10.43)

2. Secondary Outcome: Clinical Global Impression of Severity (CGI-S) Change From Baseline
Description: The CGI-S (range 1-7) is a standardized, clinician-rated assessment to rate the severity of illness of the patient. The clinician assessed the severity of illness using the following categories: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = among the most extremely ill. The minimum score is 1 and maximum score is 7, with higher scores indicating more severe illness.
Time Frame: Day 1 - Day 62
Population: Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Study Treatment
Number analyzed (Participants) | 79
Scores on a scale
  Day 13 (n=78) | -0.1 (0.39)
  Day 27 Paliperidone ER Baseline (n=79) | -0.1 (0.37)
  Day 48 (n=74) | -0.3 (0.60)
  Day 62 (n=77) | -0.4 (0.65)
  Post Day 27 Endpoint (n=79) | -0.4 (0.67)

3. Secondary Outcome: Personal and Social Performance Score (PSP) Change From Baseline
Description: The PSP (range 1-100) is a validated clinician-rated assessment of functioning. Four areas of functioning (socially useful activities, personal/social relationships, self-care, disturbing/aggressive behaviors) are assessed on a 6-point scale (0=absent to 5=very severe). A transformed score from 1 to 100 is generated from the raw score based on the clinical interpretation of the scores generated in the 4 areas of functioning, with a higher transformed score indicating better function.
Time Frame: Day 1 - Day 62
Population: Includes participants in the efficacy analysis set for with PSP scores available.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Study Treatment
Number analyzed (Participants) | 78
Scores on a scale
  Day 27 Paliperidone ER Baseline (n=78) | 1.2 (7.25)
  Day 62 (n=76) | 2.8 (7.23)

4. Primary Outcome: The Difference in the Incidence of Any Adverse Events When Patients Switch Their Antipsychotic From Treatment as Usual (TAU) to Paliperidone ER
Description: Adverse Event summary for both serious adverse events and other adverse events. Please see the Clinical Study Report Synopsis for results on this primary outcome measure or the AE section for a detailed breakdown of each adverse event preferred term in both categories.
Time Frame: Day 1 - Day 62
Population: Safety Analysis Set
Measure: Number; unit: Participants
Groups:
- TAU Phase: Day 1 through Day 27 (4 weeks)
- Paliperidone ER Phase: Day 28 through Day 62 (1 week cross titration plus 4 weeks mono-therapy).
Arm/Group | TAU Phase | Paliperidone ER Phase
Number analyzed (Participants) | 84 | 84
Participants
  Serious Adverse Events | 0 | 2
  Other Adverse Events | 27 | 43

ADVERSE EVENTS:
Description: This was a single-arm crossover study. Data are provided for 3 groups: Treatment As Usual (TAU) - Pali ER (participants who completed Phase 1 and went on to receive study drug in Phase 2; n=84), Paliperidone ER (Phase 2; n=84), and TAU - All enrolled participants; N=114).
Groups:
- TAU - Pali ER: Phase 1; Day 1 through Day 27: Patients took therapy for schizophrenia as prescribed before study entry (referred to "treatment as usual" abbreviated as "TAU") for 4 weeks who went on to participate in Phase 2 (Paliperidone ER Phase).
- Paliperidone ER Phase: Phase 2; Day 28 through Day 62: The dose of TAU was then tapered (reduced and stopped) over a 1-week period and treatment started with paliperidone extended-release (ER) tablets, 6 mg, orally (by mouth) once daily followed by 4 weeks of paliperidone ER, 3-12 mg once daily as monotherapy (treatment with Paliperidone ER alone).
- TAU - All Enrolled Participants: Phase 1; Day 1 through Day 27: Patients took therapy for schizophrenia as prescribed before study entry (referred to "treatment as usual" abbreviated as "TAU") for 4 weeks. Phase 2; Day 28 through Day 62: The dose of TAU was then tapered (reduced and stopped) over a 1-week period and treatment started with paliperidone extended-release (ER) tablets, 6 mg, orally (by mouth) once daily followed by 4 weeks of paliperidone ER, 3-12 mg once daily as monotherapy (treatment with Paliperidone ER alone).
Arm/Group | TAU - Pali ER | Paliperidone ER Phase | TAU - All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 0/84 | 2/84 | 2/114
Other Adverse Events (participants affected / at risk) | 27/84 | 43/84 | 32/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAU - Pali ER (N=84) | Paliperidone ER Phase (N=84) | TAU - All Enrolled Participants (N=114)
Dystonia (Nervous system disorders) | 0 | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAU - Pali ER (N=84) | Paliperidone ER Phase (N=84) | TAU - All Enrolled Participants (N=114)
Vision Blurred (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Facial Pain (General disorders) | 0 | 1 | 1
Hernia Pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 2
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood Pressure Increased (Investigations) | 1 | 3 | 1
Blood Prolactin Increased (Investigations) | 1 | 3 | 1
Weight Increased (Investigations) | 5 | 3 | 5
Weight Decreased (Investigations) | 0 | 1 | 0
Increased Appetite (Metabolism and nutrition disorders) | 0 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 2 | 7 | 2
Headache (Nervous system disorders) | 3 | 6 | 3
Somnolence (Nervous system disorders) | 0 | 2 | 0
Akathisia (Nervous system disorders) | 2 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 1 | 1
Extrapyramidal Disorder (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0
Homicidal Ideation (Psychiatric disorders) | 0 | 1 | 0
Sleep Disorder (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 1 | 0 | 1
Liver Disorder (Hepatobiliary disorders) | 1 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1
Back Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Neck Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood Potassium Increased (Investigations) | 1 | 0 | 1
Blood Pressure Diastolic Decreased (Investigations) | 1 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Drooling (Nervous system disorders) | 1 | 0 | 1
Thinking Abnormal (Psychiatric disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Feces discolores (Gastrointestinal disorders) | 0 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 0 | 1
Blood Potassium Decreased (Investigations) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Please see the Clinical Study Report Synopsis for results on the primary outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days